CLINICAL TRIAL: NCT01376882
Title: Behavioural and Cerebral Haemodynamic Effects of Caffeine Withdrawal and Caffeine Administration Following 2-week Maintenance or Abstinence
Brief Title: Cognitive and Cerebral Blood Flow Effects of 2-week Caffeine Abstinence or Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Crystal Haskell, Dr, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 24G4
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Cognitive Function; Mood; Cerebral Haemodynamics; Caffeine Withdrawal
Keywords: Caffeine; Withdrawal; Cognitive function; Mood; Cerebral haemodynamics
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acute withdrawal (Experimental): Chronic intervention 100 mg caffeine capsules 3 times per day for 14 days. Acute intervention of placebo capsule on day 15.
  Interventions: Dietary Supplement: Caffeine and Placebo
- Acute caffeine-independent of withdrawal (Experimental): Chronic intervention of placebo capsules 3 times per day for 14 days. Acute intervention of 100 mg caffeine capsule on day 15.
  Interventions: Dietary Supplement: Placebo and Caffeine
- Chronic abstinence (Experimental): Chronic intervention of placebo capsules 3 times per day for 14 days. Acute intervention of placebo capsule on day 15.
  Interventions: Dietary Supplement: Placebo
- Acute caffeine-in state of withdrawal (Experimental): Chronic intervention of 100 mg caffeine capsule 3 times per day for 14 days. Acute intervention of 100 mg caffeine capsule on day 15.
  Interventions: Dietary Supplement: Caffeine

INTERVENTIONS:
Dietary Supplement: Placebo — Inert placebo containing silica powder CAB-O-SIL-M-5Pharma (Pharmaceutical grade)CABOT GmbH. 1 Size 0 capsule 3 times a day for 14 days and 1 size 0 capsule on day 15.
  Arms: Chronic abstinence
Dietary Supplement: Caffeine and Placebo — 100 mg Caffeine capsules 3 times per day for 14 days and 1 size 0 capsule of inert placebo containing silica powder CAB-O-SIL-M-5Pharma (Pharmaceutical grade)CABOT GmbH on day 15.
  Arms: Acute withdrawal
Dietary Supplement: Placebo and Caffeine — Inert placebo capsules containing silica powder CAB-O-SIL-M-5Pharma (Pharmaceutical grade)CABOT GmbH, 1 Size 0 capsule 3 times a day for 14 days and a 100mg caffeine capsule on day 15.
  Arms: Acute caffeine-independent of withdrawal
Dietary Supplement: Caffeine — Capsule containing 100 mg caffeine, one 3 times a day for 14 days and then one capsule on day 15.
  Arms: Acute caffeine-in state of withdrawal

SUMMARY:
The purpose of this study is to determine the effects of 2 weeks caffeine abstinence as compared to 2 weeks caffeine maintenance (300mg per day)on cognition and mood. Cerebral blood flow effects will also be assessed in a subset of participants. The role of caffeine abstinence/maintenance in the acute effects of caffeine will also be explored.

DETAILED DESCRIPTION:
The current randomised, placebo-controlled, double-blind, parallel groups study aims to explore the behavioural effects of 2-weeks caffeine abstinence as well as establishing the role of abstinence in the effects of caffeine administration by administering caffeine or placebo to those in a state of chronic and acute abstinence. This research also aims to explore, in a subset of participants, the cerebral blood flow effects of caffeine abstinence and caffeine administration using Near Infrared Spectroscopy (NIRS). Cerebral blood flow will be measured both at rest and during performance of cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* 18 - 40 years
* Healthy
* Consume ≥ 150 mg caffeine daily
* No herbal supplements/prescription medications (excl. contraceptive pill)
* Non smoker
* Native English speaker

Exclusion Criteria:

* Diagnosis of any significant medical condition or disorder
* Any known allergy or hypersensitivity to food.
* BMI >29.9 or <18.5
* Blood pressure >139/89

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 2 weeks
  Performance is assessed using COMPASS (Computerised Mental Performance Assessment System), which presents a battery of standard cognitive tasks assessing aspects of attention and memory.

SECONDARY OUTCOMES:
Mood | 2 weeks
  Mood will be evaluated using Visual Analogue Scales administered using COMPASS.
Cerebral haemodynamic | 2 weeks
  Cerebral blood flow will be measured in a subset of participants using Near Infrared Spectroscopy (NIRS).
Sleep | 2 weeks
  Quality of sleep will be measured using the Pitsburgh Sleep Quality Index (PSQI).
Caffeine withdrawal | 2 weeks
  Symptoms of caffeine withdrawal will be measured using a Subjective and Somatic State Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- See also: COMPASS software — http://www.cognitivetesting.co.uk